CLINICAL TRIAL: NCT02114320
Title: Multicenter Study of EUS-guided Biliary Drainage Using Partially Covered With a Dedicated Introducer or Fully Covered Antimigration Metallic Stents
Brief Title: Clinical Outcomes of EUS-guided Biliary Drainage Using Partially or Fully Covered Metallic Stents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Do Hyun Park, Dr, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUS-BD-001
Record Dates: First submitted 2014-03-31; First posted 2014-04-15 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-04

CONDITIONS: Cholestasis, Extrahepatic
Keywords: Endoscopic ultrasonography; Biliary drainage; Metal stent
MeSH Terms: conditions — Cholestasis, Extrahepatic | interventions — Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS-BD-1 (Experimental): EUS-BD-1 inserts a partially covered self-expanding metallic (hybrid) stent with a dedicated introducer for EUS-BD
  Interventions: Device: EUS-BD
- EUS-BD-2 (Experimental): EUS-BD-2 inserts a fully covered self-expanding metallic stent
  Interventions: Device: EUS-BD

INTERVENTIONS:
Device: EUS-BD — EUS-guided hepaticogastrostomy (EUS-HG) will be performed in patients with hilar stricture or altered anatomy such as Roux-en-Y anastomosis, and EUS-guided choledochoduodenostomy (EUS-CD) will be performed in patients with mid to distal extrahepatic bile duct strictures. Because EUS-guided rendezvous technique can be attempted only in patients in whom the papilla is endoscopically accessible. Following bile duct puncture using a 19-gauge fine needle, one-step or graded tract dilatation will be performed. Then, finally we insert a partially or fully covered metallic stent.
  Other Names: EUS-BD-1: a partially covered self-expanding metallic (hybrid) stent with a dedicated introducer for EUS-BD; EUS-BD-2: a fully covered self-expanding metallic stent

SUMMARY:
Although endoscopic retrograde cholangiopancreatography (ERCP) is almost always successful in patients with malignant biliary obstruction, selective biliary cannulation fails in some cases and conventional ERCP may not be possible in patients with tumor invasion of the duodenum or major papilla, surgically altered anatomy (e.g., Roux-en-Y anastomosis), or complex hilar biliary strictures. In such cases, percutaneous transhepatic biliary drainage (PTBD) is an useful alternative. However, PTBD had various complications and the presence of an external drainage catheter would also have a cosmetic problem related to the external drainage and an adverse impact on quality of life (QOL) of terminally ill patients.

Since endoscopic ultrasound-guided bile duct puncture was described in 1996, sporadic case reports of EUS-guided biliary drainage (EUS-BD) suggested that it was a feasible and effective alternative in patients with failed conventional ERCP stenting. The potential benefits of EUS-BD include one-stage procedure in ERCP unit, and internal drainage for avoiding long-term external drainage in cases where external PTBD drainage catheters cannot be internalized, thus significantly improving the QOL of terminally ill patients, and possibly lower morbidity than PTBD or surgery.

Up to date, only a few case series of EUS-BD with small numbers of patients have been published, and known the feasibility and safety in terms of the incidence of procedure-related clinical outcomes.

DETAILED DESCRIPTION:
We investigated the efficacy and safety of EUS-BD using partially covered (hybrid) metallic stent with a dedicated introducer for EUS-BD, or fully covered antimigration metallic stents in malignant biliary obstruction after failed conventional ERCP as a prospective multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* malignant biliary obstruction
* Inoperable state
* age > 18 yrs
* failed primary ERCP

Exclusion Criteria:

* uncontrolled coagulopathy
* refuse to this study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Technical success rate and procedural time of EUS-BD using metallic stents | six months
  Measure the successful rate of biliary drainage using metallic stents and procedural time

SECONDARY OUTCOMES:
Complication rate of EUS-BD using metallic stents | six months
  Measure the complication rate of EUS-BD using metallic stents

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Tae Hoon Lee, Cheonan
  - Woo Hyun Paik, Ilsan